CLINICAL TRIAL: NCT01426477
Title: Veritas in Non-Bridging Ventral Hernia Repair
Acronym: VIBE
Status: Terminated | Type: Observational
Sponsor: Baxter Healthcare Corporation (Industry)
Collaborators: Synovis Surgical Innovations (Industry)
Responsible Party: Sponsor
Other Study IDs: 09-004
Record Dates: First submitted 2011-08-29; First posted 2011-08-31 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Hernia
Keywords: Ventral hernia; Abdominal wall hernia; Incisional hernia; Biologic mesh; Veritas Collagen Matrix; Veritas
MeSH Terms: conditions — Hernia; Hernia, Ventral; Hernia, Abdominal; Incisional Hernia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Veritas Collagen Matrix: Observational study of subjects who undergo open ventral hernia repair using Veritas Collagen Matrix in an underlay technique.

SUMMARY:
The main study objective is to determine the frequency of hernia recurrence following use of Veritas Collagen Matrix.

ELIGIBILITY:
Inclusion Criteria:

* Must be 18 years of age or older
* Ability to understand and read English
* Must be scheduled for open abdominal surgery for repair of primary ventral hernia or first recurrence of a ventral hernia with the Veritas Collagen Matrix using the underlay technique, with our without component separation
* Must be of ambulatory status
* Primary closure can be obtained during surgery
* Repair is such that one piece of Veritas can be used to reinforce the repair

Exclusion Criteria:

* Hernia is undetectable on physical exam
* There is evidence of existing cancer
* BMI ≥ 40
* Use of chronic immunosuppressive therapy, including steroids or cytotoxic agents
* Any condition that product labeling indicates would adversely affect participant safety, including sensitivity to bovine products

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study surgeons will recruit patients from within their own practice, or through their typical referring sources.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Hernia recurrence | 2 Years
  Recurrence will be evaluated through physical exam and/or CT scans at all study visits (30 days, 6 months, 1 year, and 2 years), or when patients present with symptoms, with primary endpoint at 2 years.

SECONDARY OUTCOMES:
Number of Medical and Surgical Complications | 2 years
  Medical and Surgical Complications, including seroma, wound infection or other concurrent infection, hematoma, fistula, ileus, skin necrosis, wound dehiscence, or any other device-related events, will be evaluated through physical exam and/or CT scans at 30 days, 6 months, 1 year, and 2 years, or when patients present with symptoms. These will be reported as total number of each complication within the total number of patients.
Change in Quality of Life | Baseline to 2 Years
  Patients will complete questionnaires regarding physical functioning including activities of daily living, work productivity, and patient comfort at various timepoints after implant at baseline, and at all follow-up visits. Outcomes will be reported in the change from baseline to 2-years.

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Mayo Clinic Department of Surgery, Jacksonville, Florida
  - Watson Clinic Center for Research, Lakeland, Florida
  - Atlanta Colon & Rectal Surgery, P.A., Atlanta, Georgia
  - Pratt Medical Center, Fredericksburg, Virginia